CLINICAL TRIAL: NCT01800500
Title: Exploring Current Smokers' Interest in Using Smokeless Tobacco Products Smokeless Tobacco Substitution for Cigarettes
Brief Title: Interest in Smokeless Tobacco Product as a Substitution for Cigarettes in Current Smokers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty accruing
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 165309; NCI-2013-00403 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-20; First posted 2013-02-27 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (fixed rate ST product prices) (Experimental): Participants purchase ST products using a fixed rate of product prices once weekly and record their consumption of ST products and cigarettes smoked daily for 3 weeks
  Interventions: Behavioral: smoking cessation intervention; Other: questionnaire administration; Other: quality-of-life assessment; Other: laboratory biomarker analysis; Other: ecigarettes
- Arm II (escalating ST product prices) (Experimental): Participants purchase ST products using escalating product prices once weekly and record their consumption of ST products and cigarettes smoked daily for 3 weeks.
  Interventions: Behavioral: smoking cessation intervention; Other: questionnaire administration; Other: quality-of-life assessment; Other: laboratory biomarker analysis; Other: ecigarettes

INTERVENTIONS:
Behavioral: smoking cessation intervention — Purchase ST products using a fixed rate of product prices
  Arms: Arm I (fixed rate ST product prices)
Behavioral: smoking cessation intervention — Purchase ST products using escalating product prices
  Arms: Arm II (escalating ST product prices)
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies
Other: ecigarettes — Purchase ST products using escalating product prices nicotine replacement therapy
  Other Names: ecigarettes, Stonewall, Ariva, Camel Snus, and Marlboro Snus,NRT
  Arms: Arm II (escalating ST product prices)
Other: ecigarettes — Purchase ST products using a fixed rate of product prices nicotine replacement therapy
  Other Names: ecigarettes, Stonewall, Ariva, Camel Snus, and Marlboro Snus, NRT
  Arms: Arm I (fixed rate ST product prices)

SUMMARY:
This randomized clinical trial studies interest in smokeless tobacco product as a substitution for cigarettes in current smokers. Use of smokeless tobacco products may help people stop smoking. Measuring use of other sources of nicotine for cigarettes under a variety of different conditions may help determine whether and how much smokers are willing to use substitutions

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Systematically vary price, availability, product type, and information about products to examine their individual and joint effects on degree of substitution of smokeless products for cigarettes.

II. Examine the impact of smokeless tobacco (ST) substitution on biomarkers of exposure (carbon monoxide [CO], cotinine).

III. Explore relationships between ST substitution and measures of mood and health related quality of life.

OUTLINE: Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants purchase ST products using a fixed rate of product prices once weekly and record their consumption of ST products and cigarettes smoked daily for 3 weeks.

ARM II: Participants purchase ST products using escalating product prices once weekly and record their consumption of ST products and cigarettes smoked daily for 3 weeks.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Must report currently smoke at least 10 cigarettes per day and been smoking for at least 1 year
* Must not be planning to quit smoking in the next 30 days, nor tried to quit in the last 30 days
* Must be able to read and speak English
* Should not concurrently using other tobacco products or nicotine medications
* Willing to try new tobacco products and substitute other brands of cigarettes
* Not current participating in any other ongoing research study
* Must be in good general health
* Medically eligible to receive nicotine replacement products (based upon the New York State [NYS] Smokers Quit line eligibility criteria)

  * No history of heart attack or stoke in last 2 weeks
  * No current use of Zyban, bupropion, Wellbutrin, or Chantix/varenicline, or other smoking cessation medication
  * No history of chest pains or angina in past month
  * No report of physician diagnosed arrhythmia/irregular heartbeat, fast heartbeat, abnormal heart rate, or use of pacemaker
  * No current report of physician diagnosed heart disease/coronary artery disease, high blood pressure (systolic blood pressure [SBP] = 160; diastolic blood pressure [DBP] = 100), stomach ulcer, diabetes, or taking pills for depression or asthma
  * No self-reported chronic dental problems that would interfere with using oral products
  * No use of an electronic cigarette (e-cigarette) in the past 30 days
  * No known sensitivity to glycerol, propylene glycol, or glycerin
* For females, not currently pregnant or breastfeeding; nor planning to become pregnant during the follow-up interval
* Prospective participants must also pass screening tests for substance use, administered at the orientation session, to be entered on study; substance use will be assessed using a Clinical Laboratory Improvement Amendments (CLIA)-waived 7-drug urine screen (detecting presence of tetrahydrocannabinol [THC], opiates, amphetamine, barbiturates, methamphetamine, phencyclidine [PCP], and lysergic acid diethylamide [LSD]); participants must test negative on all 7 to be put on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of tobacco use accounted for by ST | Up to week 5
  Tested using hierarchical linear modeling and generalized estimating equations.
Proportion of group members that replace at least 50% of baseline cigarette consumption with ST | Up to week 5
  Assessed using a Fisher's exact test.
Change in saliva cotinine | Up to week 5
  Tested using hierarchical linear modeling and generalized estimating equations.
Change in exhaled alveolar CO | Up to week 5
  Tested using hierarchical linear modeling and generalized estimating equations.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States